CLINICAL TRIAL: NCT04960423
Title: Clinical Study of Imaging and Endoplant-related Mechanical Complications After Long Segment Fixation and Fusion of Degenerative Lumbar Scoliosis (DLS)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LM2018106
Record Dates: First submitted 2021-07-04; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Degenerative Scoliosis
MeSH Terms: interventions — Gene Fusion

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Long Segment Fixation and Fusion — Long Segment Fixation and Fusion

SUMMARY:
There is a high probability of mechanical complications in patients with degenerative lumbar scoliosis after long segment fixation and fusion, and there are few studies on distal borderline kyphosis deformity/failure. This study was designed to retrospectively analyze the patients with degenerative lumbar scoliosis (DLS) who underwent posterior selective decompression and long segment fixation and fusion surgery in the lumbar spine department of our hospital from April 2009 to May 2016. Patients' basic data, surgical data and preoperative, immediate postoperative and follow-up imaging data were collected to study the incidence of distal mechanical complications, risk factors and their relationship with clinical symptom scores in DLS patients undergoing posterior selective decompression and long segment fixation and fusion. It has guiding significance for clinical operation decision making.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥45 years old;
* The number of fixed vertebral bodies ≥5, and the upper instrumented vertebra (UIV) is located in the thoracolumbar segment;
* Third generation total pedicle screw internal fixation system;
* Follow-up time ≥24 months;
* Complete clinical and imaging data.

Exclusion Criteria:

* Idiopathic scoliosis, neuromuscular scoliosis, non-structural scoliosis, spinal tumors, spinal tuberculosis, ankylosing spondylitis, humman's disease, history of spinal surgery, history of spinal trauma, and history of hip surgery

Ages: 40 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: From April 2009 to May 2019, patients with degenerative lumbar scoliosis (DLS) underwent posterior selective decompression and long segment fixation and fusion surgery in the Department of Orthopaedic Lumbar Surgery of our hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Imaging and Endoplant-related Mechanical Complications | 2019.1.1-2025.12.31
  PJK, DJK

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University of Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No